CLINICAL TRIAL: NCT03853408
Title: Short Term Outcomes of Acute Cholecystitis Managed at a University Hospital
Status: Completed | Type: Observational
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Munirah Fetaini, Principal Investigator, King Abdulaziz University
Other Study IDs: D/39/3441
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Acute Cholecystitis
Keywords: Acute cholecystitis; Cholecystectomy; overweight; BMI; early; delayed
MeSH Terms: conditions — Cholecystitis, Acute; Overweight | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First Admission: Cholecystectomy during first admission
  Interventions: Procedure: Cholecystectomy
- Second Admission: Cholecystectomy during second admission
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Cholecystectomy (removal of the gallbladder) for acute cholecystitis

SUMMARY:
The aim of this retrospective study was to assess the different outcomes of early (performed on the patient's first admission for acute cholecystitis) and delayed cholecystectomy (done on a second admission) at King Abdulaziz University Hospital in Jeddah, Saudi Arabia.

DETAILED DESCRIPTION:
This study was conducted retrospectively through reviewing patients medical records

ELIGIBILITY:
Inclusion Criteria:

Male and female patients who presented to the Emergency Department of KAUH with an acute cholecystitis

Exclusion Criteria:

* Patients with no acute cholecystitis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data were collected retrospectively from the electronic medical records data system at KAUH. We included all adult patients who presented to the Emergency Department of KAUH with an acute cholecystitis between January 2010 and April 2018
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Type of surgery | Intraoperative (during surgery) - surgery takes an hour on an average
  Laparoscopic cholecystectomy or Laparoscopic cholecystectomy converted to open
Blood Transfusion need | Intraoperative (during surgery) - surgery takes an hour on an average
  * Yes
  * No
ICU admission: | Post operation "after surgery" immediately
  * Yes
  * No
Duration of Surgery | minutes "intraoperative" (surgery takes 1 hour on an average)
  How many minutes did the surgery take (range)
Time to operation room (hours) | hours pre surgery
  How many hours from admission to surgery
Length of stay after surgery | Days ( usually 2 days on an average )
  How many days did patients stay after surgery (range)

CONTACTS AND LOCATIONS:
Locations (1):
- King Abulaziz University, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and analyzed during this study are available upon request